CLINICAL TRIAL: NCT06871059
Title: Effectiveness, Implementation and Spillover Effects of a Culturally Adapted Diabetes Prevention Program in Spanish Primary Care Centers: a Cluster Randomized Hybrid Type II Trial
Brief Title: Effectiveness, Implementation and Spillover Effects of a Culturally Adapted DPP in Spanish Primary Care Centers
Acronym: ALADIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI23/01625
Record Dates: First submitted 2025-02-28; First posted 2025-03-11 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Prediabetes
Keywords: Diabetes Prevention Program; Prediabetes; Type 2 diabetes; Lifestyle; Disease prevention; Diet; Physical activity
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adapted Diabetes Prevention Program (Experimental): 12-month group-based behavioural program on lifestyle changes
  Interventions: Behavioral: Adapted Diabetes Prevention Program
- Usual care (Active Comparator): Usual care according to national guidelines
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Adapted Diabetes Prevention Program — Participants assigned to this group will participate in a group-based behavioural change program to improve diet and increase physical activity levels during 12 months.
  Arms: Adapted Diabetes Prevention Program
Behavioral: Usual Care — Participants assigned to this groups will receive usual care according to national guidelines
  Arms: Usual care

SUMMARY:
The ALADIM trial is a hybrid type II effectiveness-implementation cluster-randomized controlled, parallel, two arm, superiority trial. The clusters consist of 10 Primary Care Centers (PCCs) of Mallorca (Balearic Islands, Spain), which are randomly assigned to either the intervention or the control group in a 1:1 ratio. The intervention group (5 PCCs) receives training and supporting material to facilitate the implementation of the adapted DPP and effectively deliver the program over a 12-month period. The control group (5 PCCs) continues providing usual care, in line with standard healthcare practices. Effectiveness outcomes are assessed at participant level according to a cluster-randomized controlled design with data collection at baseline, 6-month and 12-month during the intervention period, and at 18-month follow-up to evaluate mid-term effects post-intervention. Implementation outcomes are assessed at PCC level throughout the study period. Prior to the hybrid trial, the DPP will be culturally and contextually adapted to the Spanish Primary Care setting.

The DPP will be culturally adapted using the Intervention Mapping ADAPT (IM-ADAPT) approach. Simultaneously, the implementation strategy will be designed using the Implementation Mapping approach.

DETAILED DESCRIPTION:
Alongside type 2 diabetes (T2D), prediabetes prevalence is also rising, placing a significant burden on public health systems, individuals, and their families.

Promoting a healthy lifestyle that includes regular physical activity, a healthy diet, smoking cessation, and achieving and maintaining a healthy body weight can effectively prevent or delay T2D onset. Major diabetes prevention trials, such as the Diabetes Prevention Program (DPP) in the United States, have demonstrated that intensive lifestyle interventions can significantly reduce T2D risk in individuals with prediabetes.However, despite strong evidence supporting the effectiveness of lifestyle interventions, and international guidelines recommending screening and referral of at-risk individuals, the global impact of scaling up diabetes prevention in real-world healthcare practice remains insufficient, most probably due to systemic (organization and leadership) and individual (healthcare professionals) barriers hindering effective implementation.

The ALADIM study aims to evaluate the effectiveness and implementation of an adapted DPP in Spanish Primary Care Centers (PCCs), using a hybrid type 2 approach. This approach addresses the gap between efficacy and effectiveness studies, providing clinically valid results while accelerating the translation of research into practice. The IM-ADAPT approach will guide the DPP adaptation to the Spanish Primary Care setting, while Implementation Mapping will inform the development, refinement, and evaluation of the implementation strategy.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years; body mass index (BMI) of ≥25 kg/m2 (≥23 kg/m2, if Asian); fasting plasma glucose (FPG) between 1010 and 125 mg/dL, or plasma glucose of 140 to 199 mg/dl measured 2 hours after a 75 g glucose load, or HbA1c between 5.7% and 6.4%, or with a documented history of gestational diabetes mellitus during a previous pregnancy.

Exclusion Criteria:

Previous diagnosis of type 1 or type 2 diabetes; current use of antidiabetic medications; pregnancy at time of enrollment; terminal illness; institutionalization; dementia or significant cognitive impairment; major surgery or hospitalization in the previous 3 months; presence of any medical or psychological condition limiting participation; and concomitant active participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Weight | Baseline, 6 and 12 months
  Change in body weight at 6 and 12 months versus baseline
Implementation fidelity | Throughout the implementation period (from baseline to 12 months)
  Degree to which the adapted DPP is delivered as intended.

SECONDARY OUTCOMES:
Spill-over effect | -1, 6 and 18 months
  Change in the percentage of individuals with prediabetes receiving lifestyle advice from their healthcare professional.

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Bennasar-Veny, PhD, Principal Investigator — University of the Baleric Islands
Locations (1):
- Gerència d'Atenció Primària de Mallorca, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennasar-Veny M, Abbate M, Colom-Rossello M, Capitan-Moyano L, Hernandez-Bermudez IC, Ricci-Cabello I, Yanez AM, Fernandez ME; ALADIM investigators. Impact of an adapted diabetes prevention program in a spanish primary care setting: protocol for a type II hybrid effectiveness-implementation cluster-randomized trial (ALADIM). Implement Sci. 2025 Jun 2;20(1):27. doi: 10.1186/s13012-025-01438-3. PMID 40457444